CLINICAL TRIAL: NCT02674620
Title: Randomized Controlled Trial of Aerobic Treadmill Exercise Treatment for Concussion
Brief Title: Trial of Aerobic Treadmill Exercise Treatment for Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panam Clinic (Other)
Responsible Party: Principal Investigator, Peter MacDonald, Research Director, Panam Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2015:020
Record Dates: First submitted 2016-01-25; First posted 2016-02-04 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2018-02

CONDITIONS: Concussion
MeSH Terms: conditions — Brain Concussion | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conservative (No Intervention): Standard conservative care of concussion
- Treadmill (Experimental): Aerobic exercise treatment for concussion
  Interventions: Other: Aerobic Exercise

INTERVENTIONS:
Other: Aerobic Exercise — Patients are treated with progressive exercise
  Arms: Treadmill

SUMMARY:
A post-concussion syndrome (PCS) diagnosis has historically led to a recommendation of continued mental and physical rest to minimize symptoms. However, this conservative approach does not consider the pathophysiological mechanisms and neurological subsystem dysfunction which mediate persistent signs and symptoms. Recently, developing research is recommending targeted therapies for specific post-concussion disorders (physiologic, vestibulo-ocular and cervicogenic). The Buffalo Concussion Treadmill Test (BCTT) is a graded aerobic test that has emerged as safe, reliable, and effective in distinguishing between post-concussion syndrome sub-types, quantifying physiological recovery, and guiding return to play decision making. It has been proposed that the results of a BCTT can be used to prescribe progressively intensifying whole body aerobic exercise (such as walking or biking), maintained at a sub-symptom threshold, to improve autoregulatory function with the potential to improve PCS symptoms. Positive results with BCTT have now made it the standard of care at the University of Buffalo Concussion Clinic and Pan Am Clinic during the management of sport related concussions. Despite its increased use in patients with post-concussion syndrome there is currently no data on the use of exercise treatment in the early stages of concussion recovery.

DETAILED DESCRIPTION:
This is a randomized controlled trial of sub-threshold (symptom-threshold) exercise therapy versus relative rest treatment in subjects with an acute phase concussion.

If a participant is eligible and consent has been given the neurosurgeon will conduct a Physical Activity Readiness Medical Examination (PARmed-X) and the participant will complete an exercise tolerance test on a treadmill (Visit 1) under the supervision of the neurosurgeon and exercise scientist. Using a standardized Balke protocol, participants will perform an incremental treadmill test to the point of symptom onset of exacerbation (increase of 2 points on an overall condition Likert scale). Those who achieve a peak Heart Rate (HR) > 150 bpm will be excluded from the study since they are close to full recovery. Those who achieve a HR > 120 but < 150 bpm and who cannot exercise to exhaustion (defined as a final rating of perceived exertion (RPE) < 17 on a Borg scale) will be randomly assigned to sub-threshold aerobic exercise (exercise at a HR equivalent to 80% of their HR achieved at symptom onset or exacerbation) or to relative rest. Any participant who does not achieve a HR > 120 bpm will return the following week for a repeat treadmill test (Visit 2). If they achieve a HR > 120 bpm but cannot exercise to exhaustion during Visit 2, they will be randomly assigned to sub-threshold exercise or to relative rest. This is because participants must demonstrate a level of exercise tolerance to have a reasonable sub-threshold (80% of achieved HR) exercise treatment prescription.

Participants randomized to sub-threshold aerobic exercise will be given a HR monitor and a specific HR intensity to exercise at 30 minutes per day. Participants randomized to rest will be asked to rest for 30 minutes per day (no structured physical or cognitive activity for at least 30 minutes per day and no participation in structured aerobic exercise during the entire study). After randomization, all subjects will have treadmill testing at all subsequent follow-ups with the neurosurgeon (every 1 to 2 weeks) to determine physiological recovery. All participants will be asked to document their symptom data into a form between 7-10 PM each evening (following that day's exercise for the exercise group), along with hours of work/school, and minutes of exercise.

The study end point for each subject is at recovery (as determined by a normal exercise level and an exam from the treating neurosurgeon).

Data Analysis

All statistics will be presented as mean ± SD. Data will be analyzed with a two-way analysis of variance to compare physiological variables for the exercise and rest groups over the duration of the study. Total test duration, maximum heart rate achieved and peak respiratory rate will be compared between the two groups with an independent samples t-test. A repeated measures ANOVA will be used for all questionnaire analyses. All analysis will be completed using SPSS 22 (IBM corp, Armonk, NY, USA) with an alpha level set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Must meet the diagnostic criteria of a concussion set forth by the Consensus Statement on Concussion in Sport 4th Annual Conference of Concussion in Sport, 2013 as determined by the treating neurosurgeon.
* Presence of concussion-related symptoms at the time of testing.
* Glasgow coma scale (GCS)=15
* Patients for who parental consent can be obtained.

Exclusion Criteria:

* Patients with a history of moderate or severe traumatic brain injury, epilepsy, or stroke.
* Patients who have been diagnosed with a skull fracture, traumatic subarachnoid hemorrhage, subdural hematoma, epidural hematoma, intraparenchymal hemorrhage, or cerebral contusion on previous neuro-imaging studies.
* Pregnant female patients.
* GCS ≤ 14.
* Patients with contraindications to exercise testing as assessed by PARmed-X assessment.
* Patients for who parental consent can not be obtained.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2015-06; Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Number of days from injury to full recovery | From date of injury (day 0) to date of recovery of symptoms (as defined in Outcome measure) or when the patient is discharged from care, whichever came first, assessed up to 180 days post-injury
  To be considered at "Full recovery", participant must meet the following criteria - Asymptomatic at rest (PCSS score under 7), participating in full school activities (as pre-injury) without symptoms, normal neurological exam, and normal vestibulo-ocular exam

CONTACTS AND LOCATIONS:
Overall Officials: Jeff R Leiter, PhD, Principal Investigator — Pan Am Clinic
Locations (1):
- Pan Am Clinic, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Leddy JJ, Baker JG, Kozlowski K, Bisson L, Willer B. Reliability of a graded exercise test for assessing recovery from concussion. Clin J Sport Med. 2011 Mar;21(2):89-94. doi: 10.1097/JSM.0b013e3181fdc721. PMID 21358497
- [Background] Leddy JJ, Kozlowski K, Fung M, Pendergast DR, Willer B. Regulatory and autoregulatory physiological dysfunction as a primary characteristic of post concussion syndrome: implications for treatment. NeuroRehabilitation. 2007;22(3):199-205. PMID 17917170